CLINICAL TRIAL: NCT00574626
Title: Randomized Trial Comparing Autologous Peripheral Blood Stem Cell Transplantation to Bone Marrow Transplantation for Patients Receiving High-Dose Chemotherapy and Transplantation for Recurrent Non-Hodgkin's Lymphoma
Brief Title: Comparing Autologous Peripheral Blood Stem Cell to Bone Marrow Transplantation for Recurrent Non-Hodgkin's Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0123-92-FB
Record Dates: First submitted 2007-12-12; First posted 2007-12-17 (Estimated); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Lymphoma
Keywords: NHL; Non Hodgkins Lymphoma; BMT; Bone Marrow Transplant; PBSCT; Peripheral Blood Stem Cell Transplant; PSCT
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin | interventions — Bone Marrow Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peripheral Blood Stem Cell Transplant (Experimental): Peripheral Blood Stem Cell Transplant
  Interventions: Procedure: PBSCT
- Bone Marrow Transplantation (Active Comparator): Bone Marrow Transplantation
  Interventions: Procedure: Bone Marrow Transplant

INTERVENTIONS:
Procedure: PBSCT — Peripheral Blood Stem Cell Transplant
  Arms: Peripheral Blood Stem Cell Transplant
Procedure: Bone Marrow Transplant — Bone Marrow Transplant
  Arms: Bone Marrow Transplantation

SUMMARY:
The purpose of this study is to evaluate the difference in relapse rates and long term event free survival in patients with intermediate grade or immunoblastic non-Hodgkin's lymphoma (NHL) whose marrow is not obviously involved with NHL who are randomized to receive either an autologous bone marrow (ABMT) or peripheral stem cell transplant (PSCT). All patients with intermediate grade NHL with histologic negative bone marrow who would otherwise meet all eligibility criteria for high-dose therapy and ABMT are eligible for this study. Patients who are eligible will be randomized to either PSCT or ABMT at the time of enrollment into our transplant program.

DETAILED DESCRIPTION:
These patients would be enrolled in a high-dose protocol using carmustine, etoposide, cytarabine, and cytoxan (BEAC) with autologous hematopoietic rescue. The patients will be stratified according to good and poor prognosis category and relapsed vs. first partial response categories. The patients will have bone marrow or peripheral stem cells collected according to standard protocols. A standardized hematopoietic growth factor will be used for mobilization and post-transplant. The patients' PSC or bone marrow (BM) product will be assayed via invitro-culture techniques for occult tumor, and by molecular biologic assays. The patients' outcome for transplantation will be evaluated with response to transplantation, relapse rates and event free survival being the measured end points.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-65
* Intermediate grade non-Hodgkin's lymphoma (International Working Formulation - Follicular large cell, Diffuse Small Cleaved, Diffuse Mixed, Diffuse Large Cell, and Immunoblastic) with histologic negative bone marrow who would otherwise meet all eligibility criteria for high-dose therapy and ABMT. These criteria are in each specific high-dose therapy protocol (i.e. Karnofsky performance status > 70, adequate organ function, HIV and Hepatitis B negative, etc.). These patients would be enrolled in a high-dose protocol using carmustine, etoposide, cytarabine, and cytoxan (BEAC) with autologous hematopoietic rescue.

Exclusion Criteria:

* Patients with bone marrow histologically involved with tumor or with a bone marrow abnormality making bone marrow harvest not possible.
* Patients whose tumor is rapidly growing which may preclude the extra time involved with the PSC collection process.
* Patients who do not otherwise meet high-dose therapy and transplantation entry criteria.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 1991-12-12 (Actual); Primary Completion 2010-05-05 (Actual); Study Completion 2010-05-05 (Actual)

PRIMARY OUTCOMES:
New Blood Cell Production Response | From date of transplant until death (up to 220 months)
  Production of new blood cells after transplantation
Percentage of Participants with Relapse | From date of transplant until death (up to 220 months)
  Percentage of participants with recurrence (return of cancer)
Percentage of participants with event free survival | From date of transplant until death (up to 220 months)
  Percentage of participants with event free survival (no relapse or progression)

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Vose, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States